CLINICAL TRIAL: NCT06634524
Title: The Effect of Dexmedetomidine on Gastric Emptying, Assessed by Ultrasound, in Patients Undergoing Laparoscopic Cholecystectomy: A Prospective Randomized Trial.
Brief Title: Effect of Dexmedetomidine on Gastric Emptying, Assessed by Ultrasound in Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Noran Hesham Mohammed Elsaid Borg, Resident of Anesthesia, Surgical Intensive Care and Pain Management, Faculty of Medicine, Tanta University, Tanta, Egypt, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264MS663/8/24
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Dexmedetomidine; Gastric Emptying; Ultrasound; Laparoscopic Cholecystectomy
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmeditomidine group (Experimental): Patients who will receive IV infusion of (0.2 µg/kg/hr dexmeditomidine).
  Interventions: Drug: Dexmeditomidine
- Control group (Placebo Comparator): Patients who will receive IV infusion of normal saline, at the same rate of dexmedetomidine infusion
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexmeditomidine — Patients who will receive IV infusion of (0.2 µg/kg/hr dexmeditomidine).
  Other Names: Group D
  Arms: Dexmeditomidine group
Drug: Normal saline — Patients who will receive IV infusion of normal saline, at the same rate of dexmedetomidine infusion.
  Other Names: Group C
  Arms: Control group

SUMMARY:
The aim of this study is to evaluate the effect of dexmedetomidine on gastric emptying assessed by gastric ultrasound in patients undergoing laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Delayed return of normal gastrointestinal function, and postoperative nausea and vomiting (PONV) are common adverse events of laparoscopic cholecystectomy under general anesthesia. Sympathetic stimulation, intra-abdominal carbon dioxide insufflation, and the consequent visceral peritoneal irritation are all contributing factors. In addition, anesthetic agents and opioids can also have a harmful impact on gastric emptying.

Dexmedetomidine, a potent and highly selective alpha-2 adrenoreceptor agonist, is frequently employed as an anesthetic adjunct in surgical procedures. By reducing the surgical stress response through its central sympatholytic and anti-inflammatory effects, dexmedetomidine offers distinct organ protection. Furthermore, its opioid-sparing effect reduces the need for perioperative analgesics.

A recent meta-analysis reported a positive impact of perioperative dexmedetomidine use on postoperative gastrointestinal function by shortening the time to pass flatus.The use of gastric ultrasound to assess cross-sectional area of the stomach and it's volume may provide better insight into the effect of dexmedetomidine on gastrointestinal function.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 21 to 65 years old.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status I-II.
* Undergoing elective laparoscopic cholecystectomy surgery

Exclusion Criteria:

* Patient's refusal.
* Patients with abnormalities in gastrointestinal tracts (including previous esophageal or gastric surgery, tumors or stricture).
* Failure to follow preoperative fasting guidelines.
* Patients with a body mass index ≥ 35
* Patients on regular treatment of antacids or prokinetic.
* Presence of history of disease causing an increase in the incidence of delayed gastric emptying such as: diabetes mellitus, obesity or electrolyte disturbances.
* Pregnancy.
* Presence of hepatic or renal dysfunction.
* Presence of existing condition causing bradycardia such as heart block, or patients on regular calcium channel blockers or beta blockers.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-10-12 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Assessment of gastric volume with the aid of ultrasound | 3 hours postoperatively
  Gastric ultrasound will be used to measure gastric volume through cross-sectional area before induction, and 1 and 3 hours postoperatively.
  Estimated gastric volumes will be calculated using a previously validated formula: gastric volume (mL) = 27.0 + (14.6 ×CSA) - (1.28 ×Age).

SECONDARY OUTCOMES:
Measurement of cross-sectional area of gastric antrum | 3 hours postoperatively
  Gastric ultrasound will be used to measure gastric volume through cross sectional area. Gastric antrum images will be obtained using 2 - 5 MHz curvilinear probe which will be positioned in the sagittal plane of epigastric region. All imaging attempts will be carried out at 2 positions: semi-recumbent and right lateral. Images of gastric antrum will be obtained by identifying the following landmarks - left anterior lobe of the liver anteriorly, inferior vena cava and abdominal aorta posteriorly.
Gastric content assessment. | 3-hour post-operative marks in post anesthesia care unit (PACU).
  We initially will assess the nature (nil, fluid, or solid particles) of the gastric contents. An empty stomach will appear as the antrum walls juxtaposed with a "fat" appearance. The clear fluid will appear as "homogeneously hypoechoic" liquid content without residues.
  Quantitative assessment of gastric contents will be carried out by measuring the anteroposterior (AP) and craniocaudal (CC) diameters of the gastric antrum 3 times for each ultrasonographic assessment. The mean value of the 3 will be recorded. The universally accepted 2 -diameter -method will be used for the measurement of antrum cross-sectional area (CSA) because it's simple and easy to perform. It will be assessed before induction of anesthesia and at the 1-hour and 3-hour post-operative marks in post anesthesia care unit (PACU).
Relation between gastric cross-sectional area to time of passage of flatus | 24 hours postoperatively
  Time of passage of flatus will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author